CLINICAL TRIAL: NCT01303510
Title: Open, Non-randomized Trial to Assess the Immunogenicity and Safety of the 2008/2009-season Influenza Vaccine in Elderly and Young Subjects According to European Medicines Agency (EMEA) Regulations
Brief Title: A Re-licensing Study to Assess the Efficacy of Inflexal V Formulated With WHO Recommended 2008/2009 Influenza Virus Strains for the Northern Hemisphere
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INF-V-A002
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Adults from 18 to 60 years old inclusive
  Interventions: Biological: Inflexal V
- Group B (Experimental): Elderly subjects aged over 60 years
  Interventions: Biological: Inflexal V

INTERVENTIONS:
Biological: Inflexal V — Inflexal V influenza vaccine, formulated for the WHO requirements ofr the 2008-2009 season, containing per 0.5 mL dose:
  * 15 µg hemagglutinin (HA) antigen of A/Brisbane/59/2007 (H1N1)-like virus
  * 15 µg HA antigen of A/Brisbane/10/2007 (H3N2)-like virus
  * 15 µg HA antigen of B/Florida/4/2006-like virus
  Dose: intramuscular administration (M. deltoideus) of a single dose of 0.5 mL on Day 1

SUMMARY:
A study to assess whether the Northern Hemisphere 2008/2009 season influenza vaccine Inflexal V fulfills the EMEA requirements for re-registration of influenza vaccines

ELIGIBILITY:
Inclusion criteria:

* Healthy female and male adults
* Aged ≥18 to ≤60 years or >60 years on Day 1
* Written informed consent

Exclusion criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of study vaccine; oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent are excluded; inhaled or topical steroids are allowed
* Known immunodeficiency (incl. leukemia, cancer, HIV seropositivity)
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or relative or spouse of the investigator
* Suspected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research Unit AG
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in Switzerland FSFV: 09-Jul-2008 LSLV: 30-Jul-2008
Period: Overall Study
Arm/Group | Group A | Group B
Started | 55 | 56
Completed | 54 | 56
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 55 | 56 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.0) | 69.3 (5.2) | 54.4 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 29 | 31 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Safety: Incidence of Solicited Local Adverse Events
Description: Safety assessments are made by the investigator at baseline and on Day 22 as well as by the subjects themselves (in a Subject Diary) for the 4-day period immediately following vaccination
Time Frame: Days 1 to 4 inclusive, and Day 22
Population: Safety population includes all subjects who received study vaccine
Measure: Number; unit: Subjects
Arm/Group | Group A | Group B
Number analyzed (Participants) | 55 | 56
Subjects
  Ecchymosis | 1 | 1
  Erythema | 6 | 6
  Induration | 7 | 3
  Pain | 30 | 12

2. Primary Outcome: Seroconversion
Description: Seroconversion rate was defined as the proportion of subjects with ≥4-fold increase in haemagglutination inhibition (HI) antibody titer and with a titer of ≥1:40
Time Frame: Day 22 ± 2 days
Population: Intention-to-treat (ITT) and According-to-protocol (ATP) populations exclude one subject lost to follow up
Measure: Number; unit: Subjects
Arm/Group | Group A | Group B
Number analyzed (Participants) | 54 | 56
Subjects
  A/Brisbane/59/2007 | 27 | 17
  A/Uruguay/716/2007 | 32 | 43
  B/Florida/4/2006 | 34 | 20

3. Primary Outcome: Seroprotection
Description: Seroprotection rate, defined as the proportion of subjects with HI antibody titer ≥1:40
Time Frame: Day 22 ± 2 days
Population: ITT/ATP
Measure: Number; unit: Subjects
Arm/Group | Group A | Group B
Number analyzed (Participants) | 54 | 56
Subjects
  A/Brisbane/59/2007 | 52 | 39
  A/Uruguay/716/2007 | 39 | 49
  B/Florida/4/2006 | 53 | 54

4. Primary Outcome: Fold Increase in Geometric Mean Titer (GMT)
Description: GMT-fold increase - calculated as the GMT on Day 22 divided by the baseline GMT value
Time Frame: Day 22/Day 1
Population: ITT/ATP
Measure: Number; unit: Fold (ratio)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 54 | 56
Fold (ratio)
  A/Brisbane/59/2007 | 9.97 | 4.36
  A/Uruguay/716/2007 | 11.54 | 17.40
  B/Florida/4/2006 | 9.90 | 2.36

5. Secondary Outcome: Incidence of Solicited Systemic Adverse Events
Description: as for outcome 1
Time Frame: Days 1 to 4 inclusive, and Day 22
Population: Safety population
Measure: Number; unit: Subjects
Arm/Group | Group A | Group B
Number analyzed (Participants) | 54 | 56
Subjects
  Shivering | 0 | 0
  Malaise | 8 | 3

ADVERSE EVENTS:
Time Frame: Safety assessments were made by the investigator at baseline and on Day 22 (± 2 days), and by subjects themselves (Subject Diary) for the 4-day period post-vaccination. SAE surveillance extended to 6 months post-vaccination.
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 36/55 | 20/56
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=55) | Group B (N=56)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Ecchymosis (General disorders) | 1 (1) | 1 (1)
Erythema (General disorders) | 6 (6) | 6 (6)
Induration (General disorders) | 7 (7) | 3 (3)
Pain (General disorders) | 30 (30) | 12 (12)
Malaise (General disorders) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator to submit all manuscripts/abstracts to the sponsor for review at least 6 weeks before submission.